CLINICAL TRIAL: NCT02483468
Title: The Effects of Cognitive Behavioral Therapy and Transcranial Current Stimulation (tDCS) on Chronic Lower Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jeffrey Borckardt, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00036590
Record Dates: First submitted 2015-06-12; First posted 2015-06-29 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Chronic Low Back Pain; Opioid Use, Unspecified
MeSH Terms: interventions — Cognitive Behavioral Therapy; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tDCS (Experimental): Active Transcranial Direct Current Stimulation - Stimulation of the left dorsolateral prefrontal cortex with 2mA of electrical current
  Interventions: Behavioral: Cognitive Behavioral Therapy for Pain; Device: Transcranial Direct Current Stimulation
- tDCS (sham) (Sham Comparator): Inactive (sham) Transcranial Direct Current Stimulation
  Interventions: Behavioral: Cognitive Behavioral Therapy for Pain; Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Pain — Cognitive-behavioral therapy (CBT) for pain management takes an active problem-solving approach to tackling the many challenges associated with the experience of chronic pain. Rather than seeing ones self as helpless and disabled because of pain, CBT encourages individuals to take back control and re-engage in activities.
  Other Names: CBT
Device: Transcranial Direct Current Stimulation — Electrical stimulation of the prefrontal cortex using 2mA of direct current
  Other Names: tDCS
  Arms: tDCS
Device: Sham Transcranial Direct Current Stimulation — Sham stimulation of the left dorsolateral prefrontal cortex
  Other Names: Sham tDCS
  Arms: tDCS (sham)

SUMMARY:
The primary objective of this study is to evaluate the effects of cognitive-behavioral therapy in combination with transcranial direct current stimulation in (1) improving pain and functionality, (2) reducing severity of opioid use disorders, and (3) reducing impairment in associated mental health areas (e.g., depression, anxiety, PTSD, sleep). The investigators will also determine the effects of treatment on neural activity in cognitive and limbic brain regions involved in pain regulation using functional magnetic resonance imaging (fMRI), and examine its relationship to opioid use severity.

DETAILED DESCRIPTION:
As a result of sustained operations in Afghanistan and Iraq, an increasing number of U.S. military personnel and Veterans are in need of effective pain management treatment. Chronic low back pain (CLBP) is the most common pain condition among returning Veterans and is associated with high levels of opioid analgesic prescribing in VA clinics. Although opioids are effective for acute pain, they are not very effective as a long-term treatment strategy. Furthermore, opioids are associated with significantly increased risk of misuse, addiction, diversion, overdose and death. Consequently, there is a critical need for the development of alternative, effective treatments for CLBP that can be implemented in VA-based healthcare settings. The proposed study will answer critical questions regarding the ability of Transcranial Direct Current Stimulation (tDCS) to augment the effects of cognitive behavioral therapy (CBT) for pain, and elucidate possible mechanisms underlying improved outcomes. tDCS is inexpensive and highly portable, making it a very scalable tool to add to current CBT interventions within the VA healthcare system. This study has the particular advantages of building directly on positive preliminary findings among civilians and is being led by a multi-disciplinary team of experts who have successfully collaborated in the past and are uniquely qualified to implement this type of investigation. The primary objective of the proposed Stage II study is to evaluate the effects of CBT in combination with tDCS in (1) improving pain and functionality, (2) reducing severity of opioid use disorders, and (3) reducing impairment in associated mental health areas (e.g., depression, anxiety, PTSD, sleep). The investigators will also determine the effects of treatment on neural activity in cognitive and limbic brain regions involved in pain regulation using functional magnetic resonance imaging (fMRI), and examine its relationship to opioid use severity. Secondary objectives are to evaluate acute lab-based pain markers and neural correlates of improvement in chronic pain using quantitative sensory testing. In order to accomplish this the investigators are: using a manualized, evidence-based CBT intervention that is already widely-disseminated within the VA system; employing a randomized, between-groups, double-blind experimental design; and examining standardized, repeated, dependent measures of change in: (a) clinical outcomes such as pain, opioid and other substance use disorders (e.g., alcohol, illicit drugs, other prescription drugs), depression, anxiety, sleep and PTSD symptomatology; and (b) process variables such as participant satisfaction, quality of life and treatment retention. The results of this study will provide important information regarding two non-pharmacologic, evidence-based interventions (CBT and tDCS), and will help inform policies and programs to better serve the needs of U.S. military personnel, Veterans, and their families. The findings from this study may help reduce public health costs and morbidity/mortality associated with chronic pain and co-morbid prescription opiate use disorders among our nation's Veterans.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 70.
2. United States Veteran or family member of a Veteran.
3. Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of the assessment instruments.
4. Subjects must be able to comprehend English.
5. Have a chronic pain condition and ≥3months duration of pain.
6. BPI score >4/10.
7. Meet DSM-5 criteria for current (i.e., past 6 months) prescription opioid use disorder (assessed via the MINI 7.0).
8. COMM score>7.
9. Subjects may also meet criteria for a mood disorder if asymptomatic or anxiety disorders (PTSD, panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive compulsive disorder). The inclusion of subjects with affective and anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with chronic pain and prescription opioid use disorders.
10. Subjects taking psychotropic medications will be required to be maintained on a stable dose for at least four weeks before study initiation. This is because initiation or change of psychotropic medications during the course of the trial may interfere with interpretation of results.
11. Must consent to random assignment to CBT + tDCS or CBT + sham tDCS.
12. Must consent to complete all treatment and follow-up visits.
13. Must live within 100 miles of the Medical University of South Carolina.

Exclusion Criteria:

1. Subjects with symptomatic psychotic/bipolar disorder and/or deemed too high risk by the study physician
2. Subjects with current suicidal or homicidal ideation and intent.
3. Subjects with a current eating disorder (bulimia, anorexia nervosa) or with dissociative identity disorder, as they are likely to require specific time-intensive psychotherapy in addition to the proposed therapy for stabilization.
4. Subjects who would present a serious suicide risk or who are likely to require hospitalization during the course of the study.
5. Subjects enrolled in ongoing behavioral therapy for pain or substance use disorders, who are not willing to discontinue these therapies for the duration of the trial. Attendance at therapeutic activities other than study sessions will be closely monitored using the Treatment Services Review.
6. Subjects on maintenance anxiolytic, antidepressant, or mood stabilizing medications, which have been initiated during the past 4 weeks. If it is determined, based on clinical criteria, that a subject needs to be started on maintenance medications for anxiety, mood or psychotic symptoms during the course of the study, they will be discontinued from the treatment trial.
7. Subjects with organic mental syndrome.
8. Pregnant women.
9. History of seizures.
10. Implanted medical devices above the waist.
11. Latex allergy.
12. Diagnosis of Fibromyalgia.
13. History of eczema or other sensitive skin conditions.
14. Known brain tumors or lesions that intersect the area of stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Borckardt, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- tDCS (Active): Active Transcranial Direct Current Stimulation - Stimulation of the left dorsolateral prefrontal cortex with 2mA of electrical current
  Cognitive Behavioral Therapy for Pain: Cognitive-behavioral therapy (CBT) for pain management takes an active problem-solving approach to tackling the many challenges associated with the experience of chronic pain. Rather than seeing ones self as helpless and disabled because of pain, CBT encourages individuals to take back control and re-engage in activities.
  Transcranial Direct Current Stimulation: Electrical stimulation of the prefrontal cortex using 2mA of direct current
Period: Overall Study
Arm/Group | tDCS (Active) | tDCS (Sham)
Started | 65 | 51
Completed (completed defined as followed up to 3 months) | 46 | 30
Not Completed | 19 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS | tDCS (Sham) | Total
Number analyzed (Participants) | 65 | 51 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.03 (11.98) | 53.08 (10.84) | 53.05 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 53 | 42 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 59 | 46 | 105
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 18 | 41
  White | 39 | 30 | 69
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Pain
Description: Average daily pain defined by item #5 on the Brief Pain Inventory (BPI). Scale on scale of 0-10; anchored with "0-no pain" and "10- pain as bad as you can imagine."
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS (Active) | tDCS (Sham)
Number analyzed (Participants) | 46 | 30
score on a scale | 5.41 (.33) | 5.96 (.38)

2. Primary Outcome: Pain Interference
Description: Pain interference defined by the mean of items 9.a ---9.i; the measure is scored on a scale of 0--10, anchored by "0-does not interfere" and "10- completely interferes"
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS (Active) | tDCS (Sham)
Number analyzed (Participants) | 46 | 30
score on a scale | 5.00 (.39) | 5.30 (.44)

3. Primary Outcome: Pain Catastrophizing
Description: Pain catastrophizing defined by total score of 13 items pain catastrophizing scale. This measure has a total score range of 0-52 where for each item is anchored by "0-not at all" and "4-all the time." Larger total score indicates more catastrophizing.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS (Active) | tDCS (Sham)
Number analyzed (Participants) | 46 | 30
score on a scale | 20.58 (2.14) | 18.11 (2.55)

4. Secondary Outcome: Opioid Misuse
Description: Current Opioid Misuse Measure scores. 17-item Likert-type scale (For each opioid misuse risk behavior item, 0="Never and 4="Very often"). Possible range is 0 to 68. Higher scores indicate more opioid misuse concerns.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS | tDCS (Sham)
Number analyzed (Participants) | 46 | 30
score on a scale | 10.76 (9.82) | 9.80 (7.25)

5. Secondary Outcome: Psychiatric Functioning (Depression)
Description: Depression: Beck Depression Inventory-II (BDI-II): The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Possible range is 0 to 63 points. Higher scores mean more depression symptoms.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS (Active) | tDCS (Sham)
Number analyzed (Participants) | 47 | 30
score on a scale | 16.00 (12.47) | 16.87 (13.54)

6. Secondary Outcome: Psychiatric Functioning (Anxiety)
Description: Beck Anxiety Inventory (BAI): 21-item self-report inventory used to assess anxiety levels in adults and adolescents. The score range is 0-63. Higher scores mean more anxiety symptoms.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS (Active) | tDCS (Sham)
Number analyzed (Participants) | 46 | 30
score on a scale | 15.88 (12.94) | 16.38 (12.61)

7. Secondary Outcome: Psychiatric Functioning (PTSD)
Description: PTSD Checklist (PCL) 20-item self-report measure of the DSM-5 symptoms of PTSD: Score range: 0-80. Higher scores mean more post-traumatic stress symptoms.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS (Active) | tDCS (Sham)
Number analyzed (Participants) | 41 | 29
score on a scale | 21.22 (14.13) | 20.37 (14.18)

8. Secondary Outcome: Psychiatric Functioning (Sleep)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated. questionnaire which assesses sleep quality and disturbances. Range of scores: 0-21. Higher scores mean more sleep disturbance.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS (Active) | tDCS (Sham)
Number analyzed (Participants) | 8 | 13
score on a scale | 10.75 (5.8) | 11.23 (3.94)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | tDCS (Active) | tDCS (Sham)
All-Cause Mortality (participants affected / at risk) | 1/65 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/51
Other Adverse Events (participants affected / at risk) | 2/65 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS (Active) (N=65) | tDCS (Sham) (N=51)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin irritation as a result of wearing actigraphy wrist device
Car accident (Social circumstances) | 1 (1) | 0 (0) — car accident unrelated to study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT02483468/Prot_SAP_001.pdf
  • Informed Consent Form (2015-02-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT02483468/ICF_000.pdf